CLINICAL TRIAL: NCT01667445
Title: Determination of Effectiveness of Periarticular Local Infiltration When Compared to Spinal Epimorph for Analgesia in Total Knee Arthroplasty
Brief Title: Evaluation of the Use of Spinal Epimorph in Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, James Howard, Orthopaedic surgeon, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 102837
Record Dates: First submitted 2012-08-07; First posted 2012-08-17 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Post-operative Pain; Osteoarthritis
Keywords: total knee arthroplasty; epimorph; analgesia
MeSH Terms: conditions — Pain, Postoperative; Osteoarthritis; Agnosia | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- epimorph (Experimental): single dose administration of 150mcg epimorph
  Interventions: Drug: Epimorph
- spinal analgesia (Active Comparator): spinal alone
  Interventions: Drug: Spinal analgesia

INTERVENTIONS:
Drug: Epimorph — Patient to receive 150ug of Epimorph with Spinal anaesthetic. Injection Cocktail includes: 10mg Morphine, 30mg Ketorolac, 3.5ug/ml (385ug total) of Ropivicaine, 2.5ug /ml (275ug total) Epinephrine with the remainder of the solution made of Normal Saline to a total volume of 110ml.
  Other Names: morphine sulfate; Duramorph PF; MS Contin; Roxano
  Arms: epimorph
Drug: Spinal analgesia — Patient to receive only Spinal anaesthetic (NO EPIMORPH). Injection Cocktail includes: 10mg Morphine, 30mg Ketorolac, 3.5ug/ml (385ug total) of Ropivicaine, 2.5ug /ml (275ug total) Epinephrine with the remainder of the solution made of Normal Saline to a total volume of 110ml.
  Other Names: Analgesia cocktail
  Arms: spinal analgesia

SUMMARY:
The purpose of this study is to determine the contribution of spinal epimorph to patient's perioperative pain management in Total Knee Arthroplasty (TKA). This study is designed to determine whether spinal epimorph and its associated complications is a necessary addition to provide adequate analgesia given the multimodal approach to pain management. It is hypothesized that perioperative local infiltration with a cocktail of local and systemic analgesics will provide equal analgesia to patients who are given both local infiltration and spinal epimorph perioperatively.

DETAILED DESCRIPTION:
This will be a randomized control trial comparing two patient populations obtained from patients who will receive a primary total knee arthroplasty at LHSC University Campus. Patient participants will be recruited and consented from the arthroplasty clinic and from the preadmit clinic at University Hospital. Both the patients and those measuring the primary outcome, namely, visual pain scales will be blinded to the experimental treatment received.

Patients will be randomized to receive either a spinal with epimorph (150ug) or a spinal with no epimorph at the time of their total hip arthroplasty. This is determined as a result of a computer generated randomization within blocks of 10 (every 10 patients there will be an even number of patients within each group). As each patient signs up they are given a consecutive study number which will determine which group they are assigned to. Note should be made that at the current time patients undergoing total joint arthroplasty may or may not receive epimorph preoperatively depending on their anaesthesiologist (personal communication with Sue Ganapathy) and so both treatment arms represent the current standard of care at LHSC. Again, spinal epimorph is currently being administered for total joint replacement, irregardless of whether or not this study is being done. It is an acceptable standard of care analgesic that is available to each anesthetist should they choose to use it. Many choose to use it as they feel it improves analgesia in patients undergoing total joint arthroplasty, which are recognized as very painful procedures (especially total knees). This is no different that one anesthetist preferring to use dilaudid for pain control and another choosing to use morphine. Both are within accepted standard of care guidelines and it is up to the individual staff to utilize the drug they feel is most beneficial. This decision is based on each individual consultant's interpretation of the available literature as well as their personal practice experience. I hope this justifies our study as we are not introducing any new treatment. Patients will receive spinal epimorph whether or not we conduct this study. As such, no formal study discontinuation rules are applicable. Both patient groups will receive medical treatment as required around the time of their procedure.

Both groups of patients will receive standardized preoperative analgesia including gabapentin (600mg), acetaminophen (975 mg) and naprosyn (500mg). Both groups will receive local anaesthesia in the form of local infiltration of the wound with a previously studied cocktail of morphine, ketoralac, epinephrine and ropivicaine. (3) Post operatively patients will remain on PCA until post operative day one and then will be changed to a standardized oral protocol including long and short acting narcotics on a PRN basis, acetaminophen (975 mg Q6h x 48hrs and then on a PRN basis), naproxyn (500mg BID x 7 days) and gabapentin (300mg BID x 7 days).

Postoperatively visual analogue pain scales will be recorded at 6, 12, 18, 24, 36 and 48hrs as well as at 1 week. Foley usage, oxygen usage, nausea/vomiting and use of antiemetics and antipruritics will also be carefully documented. Both patient groups will receive the standard post operative physiotherapy and will be discharged home with a prescription for the narcotic or analgesics that were providing them with suitable analgesia during their hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients must receive a primary total knee arthroplasty

Exclusion Criteria:

* Inability to have a spinal anaesthetic
* Intolerance to narcotic pain medication
* Inability to use a Patient Controlled Analgesia
* Revision total knee arthroplasty

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
visual analogue scale for pain | 1 week post-operatively

SECONDARY OUTCOMES:
patient report of nausea | 48hours post-operatively
patient report of pruritus | 48hours post-operatively
catheterization requirements | 48hours post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: James L Howard, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- University Hospital, London Health Sciences Centre, London, Ontario, Canada